CLINICAL TRIAL: NCT02540551
Title: Sentinel Node in Ovarian Cancer: SONAR-2
Brief Title: Sentinel Node Detection in Ovarian Cancer
Acronym: SONAR-2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low detection of the SN in patients included so far (n=11)
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Netherlands Cancer Institute (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METC152028
Record Dates: First submitted 2015-08-07; First posted 2015-09-04 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Neoplasms; Sentinel Node
MeSH Terms: conditions — Ovarian Neoplasms | interventions — technetium Tc 99m nanocolloid; sulfan blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sentinel node procedure. (Experimental): Intervention: injection of blue dye and radioactive tracer (99mTc-nanocolloid or Nanocoll) in remains of the ovarian ligaments.
  Interventions: Procedure: Injection of radioactive tracer combined with Patent Blue

INTERVENTIONS:
Procedure: Injection of radioactive tracer combined with Patent Blue — Blue dye and the radioactive isotope will be injected in the remains of the ligamentum ovarium proprium (median side) and the ligamentum infundibulo-pelvicum (lateral side), just below the peritoneum. Four syringes containing 0,2 ml patent blue and 0,15 ml (20-MBq) radioactive isotope (99mTc-nanocolloid or Nanocoll®, GE Healthcare, Eindhoven, The Netherlands) will be given. After a 15-minute interval the radioactivity the SN(s) will be identified either by the mobile gamma-camera and /or gamma-probe and / or visually (blue dye) after opening the retroperitoneal space.
  Other Names: Nanocoll; Patent Blue

SUMMARY:
Recently the investigators have shown that the SN procedure performed through the injection of tracers into the ovarian ligaments is feasible and promising in patients with clinical early stage ovarian cancer (OC). Injection of radioactive tracers resulted in the identification of SNs in all 21 patients. Before a multicentre prospective trial can be initiated, still some questions have to be answered, especially if a SN procedure still is feasable in patients with OC through injection of the tracers in the ovarian ligaments, when the ovarian tumour has already been resected, either during the same surgical procedure (ovarian tumour resected for frozen section with a malignancy as result) or at a second surgical procedure to complete the staging procedure (by laparotomy or laparoscopy).

DETAILED DESCRIPTION:
Rationale:

As most cancers, ovarian cancer also spreads to regional lymph nodes. The concept of sentinel lymph node surgery is to see whether the cancer has spread to the very first lymph node or sentinel node (SN). If the SN does not contain cancer, then there is a high likelihood that the cancer has not spread to other lymph nodes. This means that, at least theoretically, a radical lymphadenectomy could be omitted and thus the associated morbidity. The SN technique has been proven to be effective in other cancers such as breast cancer and malignant melanoma. In the gynaecological field it has been shown to be effective in vulvar cancer. Recently the investigators have shown that the SN procedure performed through the injection of tracers into the ovarian ligaments is feasible and promising in patients with clinical early stage ovarian cancer (OC). Injection of radioactive tracers resulted in the identification of SNs in all 21 patients. Before a multicentre prospective trial can be initiated, still some questions have to be answered.

Objectives:

1. To determine whether or not a SN procedure in patients with OC is feasible through injection of the tracers in the ovarian ligaments, when the ovarian tumour has already been resected

   1. during the same surgical procedure (ovarian tumour resected for frozen section with a malignancy as result)
   2. during a second surgical procedure to complete the staging procedure (by laparotomy or laparoscopy), which becomes actual when a previously resected apparently benign ovarian tumour appears to be malignant at definite pathology.
2. To determine if blue colorization of the sentinel nodes after injection of blue dye is related to the time-interval between injection and retroperitoneal exploration?
3. To determine if the technique becomes more accurate by using a mobile gamma-camera guidance during the surgical procedure.

Study design: phase I feasibility study.

Study population: the following patients will be included:

* Patients with a high suspicion of an ovarian malignancy in whom a median laparotomy and a frozen section analysis is planned.
* Patients in whom previously an adnexal mass has been removed which appeared to be malignant, in whom a surgical staging procedure is planned.

Intervention (if applicable): Injection of blue dye and the radioactive-colloid in the ligamentum ovarium proprium and the ligamentum infundibulo-pelvicum. This will be done on the side of (suspected) malignancy.

Main study parameter:

Percentage of patients in whom it is feasible to identify SN's in case the malignant ovarian mass has already been resected.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: in case the tracer is injected with the adnexal mass still in situ, the surgery is prolonged at maximum with 20-25 minutes due to the required incubation time after injection of the blue dye and radioactive isotope. A scintigram will be performed 24 hours after the surgery to determine whether residual radioactive lymph nodes can be detected. The scintigram will only be performed if the patient is capable to be transported to the nuclear department. No extra blood samples will be taken, no extra visits, physical examinations or other tests are necessary. There is no risk of tumour dissemination by injecting the tracers in the ovarian ligaments. There is a 0.07 to 2.7% risk of an allergic reaction to the blue dye. The dose of radioactive isotope given does not give adverse side effects, either to the patients or the personnel present in the operating theatre.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a high suspicion of a malignant ovarian tumour planned for exploratory laparotomy. Only when a malignancy is confirmed by frozen section, the SNs will be removed prior to proceeding with a complete staging procedure.
* Patients in whom the ovarian malignant tumour has already been resected and a second surgical procedure is planned to complete the staging procedure including lymph nodes.
* Mentally competent to give informed consent.

Exclusion Criteria:

* Previous vascular surgery of the aorta, caval vein, and/or iliac vessels.
* Previous lymphadenectomy of lymph node sampling in the iliac or para-aortal region.
* History of a malignant lymphoma.
* History of a malignant tumour in the abdominal cavity.
* Previous allergic reaction to blue dye.
* Pregnant or lactating patients.
* An allergy for human albumin.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Number of patients (%) in which sentinel node(s) are detected after injection of blue dye and tracer in the ovarian ligaments. | During the surgical procedure

SECONDARY OUTCOMES:
Number of blue colorized sentinel nodes (%) 15, 30, 45, and 60 minutes after injection. | During the surgical procedure
  In the investigator's initial feasibility study in which the tracers were injected into the ligaments of the ovary, in only 2 out of 6 patients blue-stained SNs were detected after retroperitoneal exploration. The long interval between the injection of Blue Patent and retroperitoneal exploration of at least 50 min in this study may have caused the blue dye to fade before the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Kruitwagen, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC, Dept. Obst&Gyn, Maastricht, Netherlands

REFERENCES:
- [Result] Kleppe M, Brans B, Van Gorp T, Slangen BF, Kruse AJ, Pooters IN, Lotz MG, Van de Vijver KK, Kruitwagen RF. The detection of sentinel nodes in ovarian cancer: a feasibility study. J Nucl Med. 2014 Nov;55(11):1799-804. doi: 10.2967/jnumed.114.144329. Epub 2014 Oct 20. PMID 25332439
- [Derived] Laven P, Kruitwagen R, Zusterzeel P, Slangen B, van Gorp T, van der Pol J, Lambrechts S. Sentinel lymph node identification in early stage ovarian cancer: is it still possible after prior tumor resection? J Ovarian Res. 2021 Oct 13;14(1):132. doi: 10.1186/s13048-021-00887-w. PMID 34645514